CLINICAL TRIAL: NCT07133139
Title: Treatment Validation of an Ultrasound Imaging Biomarker for Myofascial Pain
Brief Title: Treatment Validation for Myofascial Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ajay Wasan, MD, Msc (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Ajay Wasan, MD, Msc, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY25060095; R61AT012282 (NIH)
Record Dates: First submitted 2025-08-08; First posted 2025-08-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low-back Pain (cLBP); Myofacial Pain
MeSH Terms: conditions — Facial Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Dry needling (Active Comparator)
  Interventions: Device: Dry Needling; Other: NUN Biomarker
- Sham Dry Needling (Sham Comparator)
  Interventions: Device: Sham Dry Needling; Other: NUN Biomarker

INTERVENTIONS:
Device: Dry Needling — The examiner will use the "repeated tapping" technique of Travel and Simmons in the active condition in the painful tender points and TPs. In the sham treatment, the needle tip retracts when pushed against the skin (like a ballpoint pen), and the subject feels a pointy object on their skin, which does not penetrate. Prior studies have shown that this is a credible placebo condition. Prior studies have also shown that one dry needling session is effective at least temporarily for 1-2 weeks, AND that US correlates of TPs improve as well
  Arms: Dry needling
Device: Sham Dry Needling — Half of the subjects will receive a sham needle instead which puts pressure on the skin but does not penetrate the skin (like a ballpoint pen with the tip retracted pushing on the skin). Since manual pressure over myofascial tender and trigger points is also an accepted treatment, the sham procedure could also be therapeutic, although we do not think it will be very effective.
  Arms: Sham Dry Needling
Other: NUN Biomarker — A NUN biomarker measurement means checking the level of a certain substance (the "NUN" biomarker) in your body that can give investigators clues about your condition.
  Measuring the NUN biomarker helps investigators see if a treatment is working or if your condition is changing.

SUMMARY:
The goal of this clinical trial is to see if a body test called the NUN biomarker can track changes in chronic low back pain after dry needling and predict who will feel better. This study is for adults with chronic low back pain from muscle pain (Myofacial Pain).

The main questions are:

* Does the biomarker drop when pain improves?
* Can it predict who benefits most?
* Do higher starting levels mean better results with real dry needling?

Investigators will compare real and fake (sham) dry needling using ultrasound, muscle pressure tests, and pain reports before and after treatment.

DETAILED DESCRIPTION:
The goal of this clinical trial is to see if a special body measurement biomarker (called the NUN biomarker) can show changes after dry needling treatment and if it can predict who will get the most pain relief. The study focuses on adults with chronic low back pain (cLBP) that also has a muscle pain (myofascial pain, MP) component.

The main questions it aims to answer are:

1. Does the NUN biomarker go down after dry needling when muscle pain gets better?
2. Can the biomarker predict who will feel better after treatment?
3. Do people with higher biomarker levels at the start respond better to dry needling than to a fake (sham) treatment?

Investigators will compare real dry needling to sham dry needling (fake treatment) to see if the biomarker changes more with real treatment and if this matches pain relief.

Participants will:

1. Get either real dry needling or sham dry needling in a single-blinded setup (participant won't know which one they're getting).
2. Have ultrasound imaging to measure the biomarker before and after treatment.
3. Take a pressure pain test to see how sensitive their muscles are.
4. Report their pain levels after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-70;
* Predominantly axial LBP (meeting NIH definition of cLBP with daily pain for at least 3 months) with a MP component as determined by the standardized examination for MP;
* Average pain score of > 3/10, with low back pain being the primary pain site;
* CLBP meeting Quebec Task Force Classification System categories I-III (from axial pain only to pain radiating beyond the knee without neurological signs). Constant radicular pain associated with sensory loss is likely a confounder to dry needling treatment success;
* NO HISTORY of receiving dry needling, to improve the effectiveness of the blind;
* Demonstration of healthcare seeking at some point for LBP.

Exclusion Criteria:

* Back surgery within the past six months;
* Active workers' compensation or litigation claims, since these patients are more likely to have exaggerated pain behavior;
* New pain treatments within 2 weeks of enrollment;
* Any clinically unstable systemic illness or condition that is judged to interfere with the trial;
* Non-ambulatory status;
* Not able to complete the questionnaire
* Currently pregnant or have intentions to become pregnant during the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Significant decrease in NUN biomarker levels in the dry needling treatment group compared to the sham (placebo) group. | 1 week after treatment at the 2nd scan session
  Relationships between changes in the biomarker and changes in the clinical condition
Correlations between changes in the biomarker and changes in the clinical assessment of myofascial pain: tender points, trigger points, and pressure algometry. | 1 week after treatment at the 2nd exam session
  relationships between changes in the biomarker and the quantitative measures on the structured clinical exam

SECONDARY OUTCOMES:
Average Pain Intensity | 3 days after treatment
  0-10 average pain intensity over the past 7 days. 0=no pain, 10=worst possible pain
Pain interference | 3 days after treatment
  Pain Interference T score on the PROMIS short form, range 0-100, lower score= less pain interference

CONTACTS AND LOCATIONS:
Overall Officials: Kang Kim, PhD, Principal Investigator — University of Pittsburgh; Ajay Wasan, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- Kauffman Medical Building, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset can be shared with investigators upon request
Supporting Information: Study Protocol, SAP
Time Frame: Available after publication of the primary paper